CLINICAL TRIAL: NCT07407179
Title: Quality of Life and Lymphedema After Surgical Treatment of Gynecological Malignancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Oncology Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: OI-695-GYN-QOL-2022
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Gynecologic Cancer
Keywords: Gynecologic Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical Treatment Group (Other): Patients undergoing radical surgical treatment for gynecological malignancies (endometrial, cervical, ovarian, and fallopian tube cancer) will be assessed for quality of life and lower limb lymphedema after treatment.
  Interventions: Procedure: Radical Surgical Treatment for Gynecological Malignancies

INTERVENTIONS:
Procedure: Radical Surgical Treatment for Gynecological Malignancies — Radical surgical treatment performed as standard of care for gynecological malignancies (endometrial, cervical, ovarian, and fallopian tube cancer), followed by assessment of quality of life and evaluation of lower limb lymphedema.

SUMMARY:
This prospective clinical study evaluates the accuracy of the currently used planning target volume (PTV) safety margin of 0.5 cm for stereotactic body radiotherapy (SBRT) of lung tumors at the Institute of Oncology Ljubljana. The study will assess setup errors and intrafractional motion using cone beam CT (CBCT) imaging in patients treated on three linear accelerators and with two different immobilization systems (vacuum cushion and long thermoplastic mask). Based on the collected data, the study aims to determine whether the current PTV margin is adequate and whether the SBRT setup protocol could be optimized.

DETAILED DESCRIPTION:
This is a prospective cohort study designed to evaluate setup errors and intrafractional motion in patients undergoing stereotactic body radiotherapy (SBRT) for lung tumors. SBRT is a highly precise, image-guided form of hypofractionated radiotherapy in which high radiation doses are delivered in 1-8 fractions. Due to the high daily dose per fraction, accurate patient positioning and motion management are essential.

At the Institute of Oncology Ljubljana, lung SBRT has been performed since 2016 using a standard PTV margin of 0.5 cm, based on published literature. However, setup accuracy and residual positioning errors may depend on local clinical workflow, imaging verification protocols, and characteristics of the simulation and treatment equipment. Therefore, it is necessary to evaluate institution-specific setup uncertainties and verify whether the current margin remains appropriate.

The study will include consecutive patients treated with lung SBRT on three treatment machines (Ap4, Ap6, and Ap7). Two immobilization methods will be evaluated: a vacuum cushion and a long thermoplastic mask. For each treatment fraction, CBCT imaging will be performed before treatment, after online correction (residual setup error), and after treatment delivery (intrafractional motion). Setup errors and motion data will be recorded for analysis.

The primary outcomes will be systematic and random setup errors, residual intrafractional error, and calculation of an appropriate PTV margin for each machine and immobilization method using a modified van Herk formula. The study will also evaluate whether the current clinical workflow could be safely shortened by reducing the frequency of CBCT imaging.

The results of this study may support optimization of local SBRT protocols and improve efficiency while maintaining patient safety and treatment accuracy.

ELIGIBILITY:
Inclusion Criteria:

Female patients aged ≥18 years

Diagnosed with gynecological malignancy (endometrial cancer, cervical cancer, ovarian cancer, or fallopian tube cancer)

Undergoing radical surgical treatment

Ability to complete quality-of-life questionnaires

Signed informed consent

Exclusion Criteria:

Age <18 years

Patients who do not undergo surgical treatment

Inability to complete questionnaires due to cognitive impairment or language barriers

Refusal or inability to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Quality of Life After Radical Surgical Treatment of Gynecological Malignancies | Up to 6 months after surgery
  Assessment of patient-reported quality of life after radical surgical treatment of gynecological malignancies (endometrial, cervical, ovarian, and fallopian tube cancer) using validated quality-of-life questionnaires.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Oncology Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No